CLINICAL TRIAL: NCT01319006
Title: A Randomized, Open-label, 3-period Crossover Study in Healthy Subjects to Determine the Effect of Particle Size on the Pharmacokinetics of Single Oral 100mg Doses of GSK1278863A
Brief Title: Relative Bioavailability Study for GSK1278863A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 114703
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Anaemia
Keywords: relative bioavailability
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1278863A 100mg (X90=13um) (Experimental): single dose
  Interventions: Drug: GSK1278863A
- GSK1278863A 100mg (x90=29Um) (Experimental): single dose
  Interventions: Drug: GSK1278863A
- GSK1278863 100mg (X90=41um) (Experimental): single dose
  Interventions: Drug: GSK1278863A

INTERVENTIONS:
Drug: GSK1278863A — 100mg (x90=13um), oral tablet, single-dose with 7 day wash-out
Drug: GSK1278863A — 100mg (x90=29um), oral tablet, single-dose with 7 day wash-out
Drug: GSK1278863A — 100mg (x90=41um), oral tablet, single-dose with 7 day wash-out

SUMMARY:
A randomized, open-label, 3-period crossover study.

DETAILED DESCRIPTION:
A randomized, open label, 3-period crossover study in healthy subjects. The primary objective of this study is to determine the relative bioavailability of GSK1278863A after single oral doses of 100mg GSK1278863A tablets with particle sizes of 13, 29, or 41 micrometers (um) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including: medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.
* Male subjects with female partners of child-bearing potential must agree to use contraception methods
* Body weight >=50kg and BMI within the range 19 to 29.9kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Subjects must have a normal resting blood pressure, after having rested quietly in a supine position for at least 15 minutes, defined as: >=100mm Hg systolic/60mm Hg diastolic and <=140mm Hg systolic/90mm Hg diastolic.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG (12 lead) judged by the Investigator and /or medical monitor to potentially introduce additional risk factors and/or interfere with the study procedures.
* Significant cardiac, pulmonary, metabolic, renal, hepatic, neurological, psychiatric, or gastrointestinal conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* CPK above the normal range.
* Calculated creatinine clearance: <80mL/min.
* Subjects with a pre-exisisting condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function-that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 drinks for males or >14 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of peptic ulcer disease or of chronic rectal bleeding.
* History of malignancy. Non-melanoma skin cancer that has been definitively removed is allowed.
* Subjects with a baseline medical history of proliferative diabetic retinopathy, preproliferative diabetic retinopathy, or wet age-related macular degeneration (AMD).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* History of sensitivity to any of the investigational products, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History or sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking. History or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* Consumption of >3 servings per day of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of investigational product, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02-25 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC (0-inf)) and maximum plasma concentration (Cmax) of GSK1278863A. | pre-dose to 24 hours post-dose
  To determine the relative bioavailability of GSK1278863A after single oral doses of 100 mg GSK1278863A tablets with particle sizes of 13, 29 and 41um in healthy subjects.

SECONDARY OUTCOMES:
Cmax, AUC (0-t), AUC(0-infinite), tmax, and t1/2 (as data permit) of GSK1278863A metabolites. | pre-dose to 24 hours post-dose
  To determine the relative exposures of metabolites of GSK1278863A after single oral doses of 100 mg GSK1278863A tablets with particle sizes of 13, 29 and 41um in healthy subjects.
Safety and tolerability of investigational product as assessed by clinical monitoring of vital signs (blood pressure, pulse rate), ECGs, and laboratory data, as well as reporting of adverse events. | Duration of subject study participation
  To assess the safety and tolerability of GSK1278863A after single oral doses of 100 mg GSK1278863A tablets with particle sizes of 13, 29 and 41um in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114703 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114703?search=study&search_terms=114703#rs
- Available data/document: Clinical Study Report: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114703 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register